CLINICAL TRIAL: NCT01062347
Title: Exploring the Possibility of Using Intestinal mRNA Levels of Zinc Transporter Genes, and Changes in Their Expression Levels in Response to Zinc Supplementation as a Bio-marker for Zinc Status
Brief Title: A Novel Bio-marker of Zinc Status
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Mohammad Bakhtiar Hossain, ICDDR,B
Other Study IDs: 2006-004
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2010-02

CONDITIONS: Zinc Deficiency
Keywords: To identify a new bio-marker for zinc status
MeSH Terms: interventions — Zinc

ARMS (1):
- zinc supplementation (20 mg/d, for 7 d) (Experimental)
  Interventions: Biological: Zinc

INTERVENTIONS:
Biological: Zinc

SUMMARY:
Zinc deficiency is a widespread public health problem in developing countries. The true prevalence of this condition remains uncertain because of lack of a specific, sensitive and reliable biomarker for assessment of human zinc status. The most widely used indicator for measuring zinc status is serum zinc level, which, however, is homeostatically regulated and influenced by stress and infection. To explore the possibility of using mRNA levels of zinc responsive genes as an indicator of zinc status, Cao and Cousins suggested metallothionein (MT) mRNA level in monocytes and peripheral blood mononuclear cells as an indicator of recent zinc uptake. However, the usefulness of MT mRNA is also limited because its level is influenced by other metals, such as copper, cadmium and cobalt and it is also affected by stress. Several authors have proposed that expression of zinc transporter genes might be useful markers of Zn status. Evidence shows reduction in dietary zinc content produces a marked increase in intestinal absorption and decrease in intestinal zinc losses. As zinc homeostasis is regulated in the intestine, study of the zinc transporters in this organ may provide indication of recent zinc uptake. Recently, a few studies have begun to investigate the applicability of using white blood cell zinc transporter expression as an indicator of zinc status and found that some of the transporters are zinc responsive. The primary objective of this study is to explore whether the expression of zinc responsive genes, such as zinc transporters in human intestinal mucosal cells, can be used as indicators of zinc status. The specific aims are to compare gene expression in: a) intestinal mucosal cells obtained by duodenal biopsy, b) sloughed intestinal mucosal cells isolated from feces, and c) peripheral blood mononuclear cells (PBMC) in fasting individuals who are receiving their usual diet + placebo or their usual diet + supplemental zinc (20 mg/d for 7 days). Gene expression values from intestinal mucosal cells (biopsy) will be compared between the placebo and zinc supplemented groups. Similar comparison will be done in the cells isolated from stool and PBMCs. This study will also provide an opportunity to compare the relative responsiveness of gene expression and serum zinc concentration following supplementation and to explore the kinetics of any changes in serum zinc concentration. Thus, blood samples will be obtained for measuring serum zinc concentration on two occasions prior to the interventions and at specified intervals during and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking

Exclusion Criteria:

* Suffering from diarrhea

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-07-01 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mirpur, Dhaka, Bangladesh

REFERENCES:
- See also: International Centre for Diarrheal Disease Research, Bangladesh — http://www.icddrb.org